CLINICAL TRIAL: NCT00103272
Title: A Phase I Study of PS-341 (Velcade, Bortezomib) in Combination With 17-allylamino-17-demethoxygeldanamycin (17-AAG) in Patients With Relapsed or Refractory Hematologic Malignancies
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin and Bortezomib in Treating Patients With Relapsed or Refractory Hematologic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01463; OSU 0448; NCI-6520; CDR0000409584; OSU-2004C0084; OSU-0448; U01CA076576 (NIH)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Acute Basophilic Leukemia; Adult Acute Eosinophilic Leukemia; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia | interventions — tanespimycin; Bortezomib

ARMS (1):
- Treatment (17-AAG and bortezomib) (Experimental): Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 1-6 hours on days 1, 4, 8, and 11 and bortezomib IV over 3-5 seconds on days 4, 8, and 11 of course 1 and on days 1, 4, 8, and 11 of all subsequent courses.
  Treatment repeats every 21 days for 3-12 courses provided patient is receiving clinical benefit. Patients achieving objective response may discontinue therapy to undergo stem cell transplantation.
  Interventions: Drug: tanespimycin; Drug: bortezomib

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE

SUMMARY:
This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin and bortezomib in treating patients with relapsed or refractory hematologic cancer. Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving 17-N-allylamino-17-demethoxygeldanamycin together with bortezomib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of PS-341 (Velcade, Bortezomib) in combination with 17-allyamino-17-demethoxygeldanamycin (17-AAG) in patients with relapsed or refractory acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL).

II. To determine the MTD of PS-341 in combination with 17-AAG in patients with relapsed or refractory chronic lymphocytic leukemia (CLL), and non-Hodgkin's lymphoma (NHL).

III. To define the specific toxicities and the dose limiting toxicity (DLT) of PS-341 in combination with 17-AAG in the treatment of patients with relapsed or refractory hematologic malignancies.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics of 17-AAG alone and in combination with PS-341 in patients with AML, ALL, CLL, and NHL.

II. To evaluate 20S proteasome inhibition following combination therapy with 17-AAG and PS-341 in patients with AML, ALL, CLL, and NHL.

III. To assess the relationship between FLT3 mutational status and leukemic cell response to PS-341 and 17-AAG in patients with AML.

IV. To assess the relationship between Bcl-2 over-expression and response to 17-AAG and PS-341 in patients with AML and NHL.

V. To evaluate the effects of the combination of PS-341 and 17-AAG on Hsp90 and NF-kappaB and their downstream targets including Hsp70, Akt, phosphorylated Akt, p21, and caspases 3 and 9 in patient-derived primary AML and NHL cells.

OUTLINE: This is a dose-escalation study. Patients are stratified according to diagnosis (acute myeloid leukemia [AML] or acute lymphoblastic leukemia vs chronic lymphoctyic leukemia or non-Hodgkin's lymphoma [NHL]).

Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) intravenously (IV) over 1-6 hours on days 1, 4, 8, and 11 and bortezomib IV over 3-5 seconds on days 4, 8, and 11 of course 1 and on days 1, 4, 8, and 11 of all subsequent courses.

Treatment repeats every 21 days for 3-12 courses provided patient is receiving clinical benefit. Patients achieving objective response may discontinue therapy to undergo stem cell transplantation.Cohorts of 3-6 patients with receive escalating doses of 17-AAG and bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After the MTD is determined, an additional 20 patients (10 per stratum with AML or follicular NHL) are enrolled and receive 17-AAG and bortezomib as above at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of 1 of the following hematologic malignancies:

  * Acute myeloid leukemia or acute lymphoblastic leukemia

    * Not a candidate for potentially curative therapy
    * WBC ≤ 10,000/mm^3 OR WBC ≤ 40,000/mm^3 that is stable for 5 days (hydroxyurea allowed)
    * No acute promyelocytic leukemia
  * Non-Hodgkin's lymphoma (NHL), including 1 of the following subtypes:

    * Small lymphocytic lymphoma
    * Marginal zone lymphoma
    * Lymphoplasmacytic lymphoma
    * Follicular lymphoma
    * Mantle cell lymphoma
    * Diffuse large B-cell lymphoma
    * Anaplastic large cell lymphoma
    * Peripheral T-cell lymphoma
    * Extranodal NK/T cell lymphoma (nasal and nasal type)
    * Enteropathy-type T-cell lymphoma
    * Hepatosplenic T-cell lymphoma
    * Angioimmunoblastic T-cell lymphoma
    * Subcutaneous panniculitis-like T-cell lymphoma
  * Chronic lymphocytic leukemia (CLL)
* Patients with NHL or CLL must meet the following criteria:

  * Ineligible for, or refused potentially curative stem cell transplantation
  * Transformed lymphoma/Richter's transformation, defined as the transformation of low-grade lymphoma, including follicular lymphoma, CLL, or small lymphocytic lymphoma to high-grade lymphoma (i.e., diffuse large cell lymphoma) allowed at time of transformation
  * Evidence of ≥ 50% bone marrow involvement at the time of enrollment OR tumor tissue accessible for biopsy (for patients enrolled after the maximum tolerated dose [MTD] is determined)
  * Absolute neutrophil count ≥ 1,000/mm^3
  * Platelet count ≥ 100,000/mm^3
* Relapsed or refractory disease
* Willing to undergo serial bone marrow biopsy (for patients enrolled after the MTD is determined)
* No untreated or active CNS leukemia or lymphoma
* Performance status - ECOG 0-2
* At least 12 weeks
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine ≤ 2.0 mg/dL
* No uncontrolled cardiac disease
* No New York Heart Association class III-IV symptomatic congestive heart failure
* No unstable angina pectoris
* No serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation > 3 beats in a row) within the past 6 months
* No other uncontrolled cardiac arrhythmia or requiring antiarrhythmic drugs
* No myocardial infarction within the past year
* No active ischemic heart disease within the past year
* No congenital long QT syndrome
* No left bundle branch block
* QTc ≥ 450 msec (for men) or 470 (for women) on ECG/EKG
* No history of LVEF < 50% by MUGA or echocardiogram
* Resting ejection fraction ≥ 50% by MUGA or echocardiogram
* No prior history of cardiac toxicity after receiving anthracycline therapy (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, or mitoxantrone hydrochloride)
* No uncontrolled pulmonary disease
* No symptomatic pulmonary disease requiring oxygen or medications
* DLCO (i.e., oxygen diffusion capacity) ≥ 80% on pulmonary function testing
* Resting and exercise oxygen saturation ≥ 90% by pulse oximetry
* No ongoing pulmonary symptoms ≥ grade 2 including any of the following:

  * Dyspnea on or off exertion
  * Paroxysmal nocturnal dyspnea
  * Significant pulmonary disease including chronic obstructive or restrictive pulmonary disease
  * No prior history of pulmonary toxicity after bleomycin or carmustine
* No Medicare requirement for home oxygen (e.g., Resting O_2 saturation ≥ 90% or desaturation to ≥ 90% with exertion)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No preexisting sensory or motor peripheral neuropathy ≥ grade 2
* No history of allergic reaction to eggs
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* Prior stem cell transplantation for relapsed or refractory disease allowed
* At least 2 weeks since prior immunotherapy and recovered
* At least 2 weeks since prior chemotherapy (excluding hydroxyurea) and recovered
* No other concurrent chemotherapy
* No concurrent routine corticosteroids except for treatment of other medical problems (e.g., pulmonary, rheumatologic, or adrenal disorders)
* At least 2 weeks since prior radiotherapy and recovered
* No prior radiotherapy that potentially included the heart in the field (e.g., mantle)
* No prior history of chest radiation
* No concurrent palliative radiotherapy
* At least 2 weeks since prior investigational therapy
* Prior bortezomib allowed
* No other concurrent commercial or investigational agents or therapies for the malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of bortezomib) in combination with 17-AAG) | Day 21
  Defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Kristie Blum, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Walker AR, Klisovic R, Johnston JS, Jiang Y, Geyer S, Kefauver C, Binkley P, Byrd JC, Grever MR, Garzon R, Phelps MA, Marcucci G, Blum KA, Blum W. Pharmacokinetics and dose escalation of the heat shock protein inhibitor 17-allyamino-17-demethoxygeldanamycin in combination with bortezomib in relapsed or refractory acute myeloid leukemia. Leuk Lymphoma. 2013 Sep;54(9):1996-2002. doi: 10.3109/10428194.2012.760733. Epub 2013 Jan 24. PMID 23256542